CLINICAL TRIAL: NCT03260764
Title: the Comparison of Multifocal Contact Lenses and Bifocal Spectacles for Congenital Cataracts
Brief Title: Multifocal Contact Lenses vs Bifocal Spectacles for Congenital Cataracts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCPMOH2017-China-7
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Multifocal Contact Lenses
Keywords: Multifocal Contact Lenses; Bifocal Spectacles; Congenital Cataracts

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group A (Experimental)
  Interventions: Device: short term Multifocal Contact Lenses; Device: short term Bifocal Spectacles
- group B (Placebo Comparator)
  Interventions: Device: short term Multifocal Contact Lenses; Device: short term Bifocal Spectacles
- group C (Experimental)
  Interventions: Device: long term Multifocal Contact Lenses
- group D (Placebo Comparator)
  Interventions: Device: long term Bifocal Spectacles

INTERVENTIONS:
Device: short term Multifocal Contact Lenses — wearing Multifocal Contact Lenses for one week
  Arms: group A; group B
Device: short term Bifocal Spectacles — wearing Bifocal Spectacles for one week
  Arms: group A; group B
Device: long term Multifocal Contact Lenses — wearing Multifocal Contact Lenses for one year
  Arms: group C
Device: long term Bifocal Spectacles — wearing Bifocal Spectacles for one year
  Arms: group D

SUMMARY:
In this study, the investigators provide participants who had congenital cataract the multifocal contact lenses and bifocal spectacles in the purpose of seeking out a better way to make a definite diagnosis with high efficiency and accuracy, and report a prospective, randomized controlled study aiming at comparison of multifocal contact lenses and bifocal spectacles.

DETAILED DESCRIPTION:
Children diagnosed as cataract without treatment were enrolled to a prospective, randomized controlled study. Patients were assigned to four groups: participants in group A wearing multifocal contact lenses a week and then bifocal spectacles a week;in Group B, the participants wearing bifocal spectacles a week and then multifocal contact lenses;in Group C, the participants wearing multifocal contact lenses four a year;in Group D, the participants wearing bifocal spectacles four a year. Investigators compare the acuity, refraction, contrast sensitivity and the results of questionnaire between A and B , C and D groups.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as binocular cataract
* after the surgery of binocular intraocular lens implantation more than one month

Exclusion Criteria:

* diagnosed as xerophthalmus
* diagnosed as other eye diseases or systemic diseases

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2017-08-20 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Demography (age, sex, laterality and medical history) | baseline
  The demography of cataract and healthy children were recorded by using a semi-structured questionnaire.

SECONDARY OUTCOMES:
The refraction status (presented as spherical equivalent, SE) | after wearing contact lenses one month, three months ,six months and a year
  Refractions were conducted with objective retinoscopy and cycloplegia, and performed by experienced optometrists
acuity | after wearing contact lenses one month, three months ,six months and a year
contrast sensitivity | after wearing contact lenses one month, three months ,six months and a year
questionnaire result | after wearing contact lenses one month, three months ,six months and a year
  the feel of wearing during different daily activities

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, M.D,Ph.D, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China